CLINICAL TRIAL: NCT02913339
Title: MHealth Interventions to Improve Access and Coverage of Uninsured People With High Cardiovascular Risk in Argentina.
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Institute for Clinical Effectiveness and Health Policy (Other)
Responsible Party: Principal Investigator, Thomas A Gaziano, Director, Global CVD Health Policy and Prevention Unit, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2015P002360
Record Dates: First submitted 2016-09-21; First posted 2016-09-23 (Estimated); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Cardiovascular Disease
Keywords: screening; telemedicine; risk assessment; prevention
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Community health workers (CHWs) will conduct screening for CVD risk using a mobile phone application to assess risk and to schedule appointments at primary care centers (PCCs). The screening process will be non-invasive and no surgical, pharmaceutical, or other testing procedures will be utilized for screening of CVD risk by CHWs. If the CHW calculates the risk of CVD to be > 10%, s/he will schedule a clinical visit with a health professional at one of the PCCs for further assessment and/or appropriate treatment. An automatic reminder messaging system will send reminder messages about upcoming appointments to the participants.
  Interventions: Other: mHealth Risk Assessment
- Control (Active Comparator): The protocol will be identical to that implemented in the intervention arm with the following difference:
  If the CHW calculates the risk of CVD to be > 10%, s/he will verbally advise the study participant of her/his increased risk and recommend that s/he schedule a clinical visit with a health professional at one of the PCCs for further assessment and/or appropriate treatment.
  Interventions: Other: mHealth Risk Assessment

INTERVENTIONS:
Other: mHealth Risk Assessment — Using mobile phone application to calculate CVD risk and to schedule interviews at local government clinics.

SUMMARY:
Cardiovascular disease (CVD) accounts for approximately one-third of Argentina's deaths. Despite the availability of management and treatment for CVD which is offered to the uninsured population at government primary care clinics (PCCs), the rates at which those at risk are screened, identified and referred to the clinics are very low. This study will determine if providing CHWs with an mHealth application using an integrated, inexpensive and validated screening tool on cell phones for screening in the community which is linked with the PCC scheduling system wirelessly allowing the CHWs to make appointments at the time they identify high-risk individuals, will increase the number of referral and follow-up visits that patients attend at the PCCs.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is a leading cause of death in Argentina where death rates have continued to rise along with risk factors for CVD. Challenges to control in low- and middle income countries (LMIC) include low awareness, shortages of trained health care workers, overcrowded primary care centers (PCCs), and overall lack of resources in health care systems. Determining ways to increase screening in community settings and efficient referral to PCCs is a significant priority in reducing the CVD burden in Argentina. Previous work funded by the NIH shows that effective low-cost screening tools are available, CHWs can be trained to use a validated, simple non-lab based screening tool in communities to identify those at high CVD risk, and use of a mobile phone application for this tool reduced both the cost of training and screening time for CHWs. What has not been shown is whether persons at high risk for CVD can be appropriately referred for proper evaluation, treatment, and effective management of CVD at the PCCs. The Ministry of Health in Argentina has instituted an incentive system through the REDES Program that has the goal of increasing the number of uninsured who are at high risk for CVD are screened, identified, referred, and provided with appropriate care and treatment with essential diagnostics and medicines. The investigators propose to develop a mHealth tool that integrates the cell phone application for the risk screening tool to be wirelessly and directly connected with the electronic scheduling systems at PCCs. This will allow CHWs to access the appointment scheduling system at the government clinics, allowing them to make appointments for the identified high-risk individuals at the time of screening to increase the number of referral and follow-up visits that these individuals attend. This integrated scheduling system will allow for text messaging to be used to remind patients of their appointments and to schedule followup care. Finally, the system will be integrated with the electronic record system at the PCC so that ongoing monitoring and evaluation of the program can be implemented. The investigators propose a pragmatic cluster randomized trial in which individual PCCs will be randomized to either to use of the integrated mHealth tool, or usual screening procedures using existing paper based screening. The objectives will be to determine if use of the mHealth tool increases the number of high-risk persons who show up for the referral visits, if it increases the rate of subsequent follow-up care visits for the referred persons, and the cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

Uninsured subjects aged 2:40 years who live in the catchment area of the participating primary care clinics with a mobile for personal use and a 10-year CVD risk of;:;: 10%, as classified by a community health worker.

Exclusion Criteria:

Pregnant women, bed-bound illiterate and persons who cannot give informed consent, or are planning to move away from the vicinity of the clinic in the following year will be excluded.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2016-08-24 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-12-29 (Actual)

PRIMARY OUTCOMES:
Impact of mHealth app on rate of uninsured persons who are at risk and attend a first visit with a health professional at a local government primary care clinic. | 6 weeks
  Proportion of patients with a 10-year CVD risk ≥ 10% that have successfully completed the baseline (first) visit to a clinic out of all those classified as having risk >10% within the prior 6 weeks in the community.

SECONDARY OUTCOMES:
Impact of mHealth app on rate of uninsured persons who are at risk and attend a follow-up visit, after baseline, with a health professional at a local government primary care clinic. | 4 months
  Proportion of patients with a 10-year CVD risk ≥ 10% that have successful completed the follow-up visit to a clinic within 4 months of the baseline visit out of all those classified as having risk >10% in the community.

OTHER OUTCOMES:
Impact of mHealth app on rate of uninsured persons who are at risk and have treatment initiated by a health professional at the government primary care clinics. | 6-12 months
  3. Proportion of patients who are on chronic medications for respective conditions and have a 5-year CVD risk ≥ 10% (i.e.Antihypertensives if systolic blood pressure (SBP)> 140 mmHg or Statins if CVD risk ≥ 20%).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Gaziano, MD, MSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- IECS- Instituto de Efectividad Clínica y Sanitaria, Buenos Aires, Buenos Aires, Argentina

REFERENCES:
- [Derived] Palmer MJ, Machiyama K, Woodd S, Gubijev A, Barnard S, Russell S, Perel P, Free C. Mobile phone-based interventions for improving adherence to medication prescribed for the primary prevention of cardiovascular disease in adults. Cochrane Database Syst Rev. 2021 Mar 26;3(3):CD012675. doi: 10.1002/14651858.CD012675.pub3. PMID 33769555
- [Derived] Beratarrechea A, Abrahams-Gessel S, Irazola V, Gutierrez L, Moyano D, Gaziano TA. Using mH ealth Tools to Improve Access and Coverage of People With Public Health Insurance and High Cardiovascular Disease Risk in Argentina: A Pragmatic Cluster Randomized Trial. J Am Heart Assoc. 2019 Apr 16;8(8):e011799. doi: 10.1161/JAHA.118.011799. PMID 30943824